CLINICAL TRIAL: NCT06498011
Title: Comparing the Effect of a Graded Repetitive Arm Supplementary Home-based Exercise Programme With COgnitive-somatoSensory-MOtor Training to Improve Arm and Hand Function After Stroke (iCOSMO)
Brief Title: COgnitive-somatoSensory-MOtor Training to Improve Arm and Hand Function After Stroke (iCOSMO)
Acronym: iCOSMO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: StrokeCog clinical training platform (Unknown)
Responsible Party: Principal Investigator, Mark Bayley, Medical Director, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22-5628
Record Dates: First submitted 2024-06-24; First posted 2024-07-12 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Stroke; CVA; Cerebrovascular Accident
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants will be blinded to the hypotheses being tested in this study i.e the participant will not be informed about the feasibility testing of the iCOSMO training intervention. The participants will also not be informed which amongst the two interventions is the experimental or control interventions, respectively. The outcome assessor will be blinded to the intervention delivered to participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iCOSMO (Experimental): 20 participants will receive the iCOSMO intervention. iCOSMO consists of two training approaches that will include active touch and movement exploratory procedures during goal-oriented tasks as well as robotic training using the Kinarm Exoskeleton device.
  Interventions: Other: integrated Somatosensory-MOtor training using a COgnitive approach(iCOSMO)
- Home GRASP (Active Comparator): 20 participants will receive the control intervention. The control group will receive a matched dose of a home-based exercise programme. The home-based exercise programme will be based on the Home Graded Repetitive Arm Supplementary Program.
  Interventions: Other: Home Graded Repetitive Arm Supplementary Program (GRASP)

INTERVENTIONS:
Other: Home Graded Repetitive Arm Supplementary Program (GRASP) — The home-based exercise programme will be based on the Home Graded Repetitive Arm Supplementary Program focusing on stretching, arm strengthening, hand strengthening, coordination and hand skills. The Home Graded Repetitive Arm Supplementary Program will be delivered 2 hours/session, 3 times/week, for 6 weeks.
  Arms: Home GRASP
Other: integrated Somatosensory-MOtor training using a COgnitive approach(iCOSMO) — The first training approach of iCOSMO will focus on integrated somatosensory-motor variables during reaching and object manipulation (60 minutes). The second training approach will focus on proprioceptive, motor and cognitive tasks using the Kinarm robotic exoskeleton (60 minutes). iCOSMO will be delivered 3 times per week (2 hours per session) for 6 weeks (Total: 36 hours of treatment).
  Arms: iCOSMO

SUMMARY:
The iCOSMO study investigates the feasibility and beneficial effects of an intervention combining sensation, motor and cognition to improve arm and hand function after chronic stroke.

DETAILED DESCRIPTION:
The iCOSMO is a two-arm randomized controlled trial study evaluating the feasibility and efficacy of combined somatosensory-motor intervention using a cognitive approach to improve upper limb recovery in people with chronic stroke. Forty participants will be recruited (20 in experimental group and 20 in the control group). iCOSMO will include active touch and movement exploratory procedures during goal-oriented tasks as well as robotic training using the Kinarm Exoskeleton device. The experimental group will receive a total of 36 hours of treatment (6 weeks). The control group will receive a matched dose of a home-based motor exercise programme. The outcome measures will include measures of feasibility such as the recruitment and adherence rates and standardised clinical and robotic assessments. The participants will be tested at the start and end of the baseline phase, at post-intervention and at 1-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stroke
* Must be more than 6 months post-stroke
* Must be above 18 years old
* Must have some motor and/or somatosensory deficits in the upper limbs

Exclusion Criteria:

* A prior history of central nervous system dysfunction other than stroke
* Upper limb deficits resulting from non-stroke pathology
* Inability to cooperate, follow instructions or provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Fidelity | Through study completion, an average of 6 weeks
  Measures of fidelity will monitor intervention delivery such as the number of intervention sessions attended and the amount of practice.
Kinarm standard tasks- the Reverse Visually Guided Reaching | Baseline, immediately after intervention,1-month
  The Kinarm standard tasks™ will include the Reverse Visually Guided Reaching. The Reverse Visually Guided Reaching task assesses attention, inhibitory control and cognitive control of visuomotor skills. A task score will be reported as a measure of a participant's performance against healthy populations.
Kinarm standard tasks- the Trail Making A&B | Baseline, immediately after intervention,1-month
  The Kinarm standard tasks™ will include the Trail Making A&B. The Trail Making tests evaluate task switching abilities. There are 2 parts of this test. Trail A: trace a sequence of targets numbered 1 to 25; Trail B: Trace alternating numeric-alpha sequence of targets 1-A-2-B etc. A task score will be reported as a measure of a participant's performance against healthy populations.
Kinarm standard tasks- the Object Hit and Avoid | Baseline, immediately after intervention,1-month
  The Kinarm standard tasks™ will include the Object Hit and Avoid. The Object Hit and Avoid task assesses spatial attention, rapid motor selection and inhibition control. A task score will be reported as a measure of a participant's performance against healthy populations.
Kinarm standard tasks- the Spatial Span Task | Baseline, immediately after intervention,1-month
  The Kinarm standard tasks™ will include the Spatial Span Task. The Spatial Span test evaluates visuospatial working memory. A task score will be reported as a measure of a participant's performance against healthy populations.
Kinarm standard tasks- the Paired Associates Learning | Baseline, immediately after intervention,1-month
  The Kinarm standard tasks™ will include the Paired Associates Learning. The Paired Associates Learning task evaluates visuospatial working memory by testing the ability to associate patterns with spatial locations and recall them after a delay. A task score will be reported as a measure of a participant's performance against healthy populations.
Kinarm standard tasks- the Visually Guided Reaching | Baseline, immediately after intervention,1-month
  The Kinarm standard tasks™ will include the Visually Guided Reaching. The Visually Guided Reaching task measures the subject's visuomotor capabilities and multi-joint coordination. A task score will reported as a measure of a participant's performance against healthy populations.
Kinarm standard tasks- the Object Hit | Baseline, immediately after intervention,1-month
  The Kinarm standard tasks™ will include the Object Hit. The Object Hit task is a rapid sensorimotor decision and control test. A task score will be reported as a measure of a participant's performance against healthy populations.
Kinarm standard tasks- the Ball-on-Bar | Baseline, immediately after intervention,1-month
  The Kinarm standard tasks™ will include the Ball-on-Bar. The Ball on Bar task assesses bimanual coordination and visuomotor skills. A task score will reported as a measure of a participant's performance against healthy populations.
Kinarm standard tasks- the Arm Posture Perturbation | Baseline, immediately after intervention,1-month
  The Kinarm standard tasks™ will include the Arm Posture Perturbation. The Arm Posture Perturbation task assesses the responsiveness to unexpected disturbances to the arm. A task score will reported as a measure of a participant's performance against healthy populations.
Kinarm standard tasks- the Arm Positioning Matching | Baseline, immediately after intervention,1-month
  The Kinarm standard tasks™ will include the Arm Positioning Matching: The Arm Position Matching task measures of a subject's proprioceptive capabilities in the upper limb. A task score will be reported as a measure of a participant's performance against healthy populations.
Kinarm standard tasks- the Arm Movement Matching | Baseline, immediately after intervention,1-month
  The Kinarm standard tasks™ will include the Arm Movement Matching: The Arm Movement Matching task assesses the ability of a subject to perceive limb motion or kinesthesia in a workspace. A task score will be reported as a measure of a participant's performance against healthy populations.
Fugl-Meyer Assessment-Upper Extremity (FMA-UE) | Baseline, immediately after intervention,1-month
  FMA-UE provides quantitative measures of sensory and motor impairments in the upper limbs and is scored from 0-66.
Action Research Arm Test (ARAT) | Baseline, immediately after intervention,1-month
  The ARAT assesses motor performance of the upper limb. It consists of 19 tasks across the 4 subscales (grasp, grip, pinch, gross movement).
Grip dynamometry | Baseline, immediately after intervention,1-month
  Maximum voluntary grip strength with the Jamar dynamometer will be used as a conventional measure of muscle strength in the upper limb post-stroke.
Pinch strength | Baseline, immediately after intervention,1-month
  Pulp-to-pulp pinch strength will be assessed using a pinch gauge (B & L Engineering).
Box and Block Test (BBT) | Baseline, immediately after intervention,1-month
  The BBT will be used to assess gross manual dexterity.

SECONDARY OUTCOMES:
Stanford Fatigue Visual Analogue Scale (SFVAS) | Through study completion, an average of 6 weeks
  The SFVAS, a single-item scale with a rating of 1 (no fatigue) to 10 (severe fatigue), will be used to assess the presence and extent of mental and physical fatigue.
Pain visual analogue scale (PVAS) | Through study completion, an average of 6 weeks
  PVAS is a single-item scale ranging from 0 (no pain) to 10 (excruciating pain).

CONTACTS AND LOCATIONS:
Overall Officials: Mark Bayley, MD, Principal Investigator — Toronto Rehabilitation Institute
Locations (1):
- Toronto Rehabilitation Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
We do not plan to share the data from this study with any researchers outside this study.

REFERENCES:
- [Background] Gopaul U, van Vliet P, Callister R, Nilsson M, Carey L. COMbined Physical and somatoSEnsory training after stroke: Development and description of a novel intervention to improve upper limb function. Physiother Res Int. 2019 Jan;24(1):e1748. doi: 10.1002/pri.1748. Epub 2018 Sep 19. PMID 30230136
- [Background] Birkenmeier RL, Prager EM, Lang CE. Translating animal doses of task-specific training to people with chronic stroke in 1-hour therapy sessions: a proof-of-concept study. Neurorehabil Neural Repair. 2010 Sep;24(7):620-35. doi: 10.1177/1545968310361957. Epub 2010 Apr 27. PMID 20424192
- [Background] Ritter PL, Gonzalez VM, Laurent DD, Lorig KR. Measurement of pain using the visual numeric scale. J Rheumatol. 2006 Mar;33(3):574-80. PMID 16511926
- [Background] Bourke TC, Lowrey CR, Dukelow SP, Bagg SD, Norman KE, Scott SH. A robot-based behavioural task to quantify impairments in rapid motor decisions and actions after stroke. J Neuroeng Rehabil. 2016 Oct 10;13(1):91. doi: 10.1186/s12984-016-0201-2. PMID 27724945
- [Background] Duncan PW, Propst M, Nelson SG. Reliability of the Fugl-Meyer assessment of sensorimotor recovery following cerebrovascular accident. Phys Ther. 1983 Oct;63(10):1606-10. doi: 10.1093/ptj/63.10.1606. PMID 6622535
- [Background] Ekstrand E, Lexell J, Brogardh C. Grip strength is a representative measure of muscle weakness in the upper extremity after stroke. Top Stroke Rehabil. 2016 Dec;23(6):400-405. doi: 10.1080/10749357.2016.1168591. Epub 2016 May 4. PMID 27145212
- [Background] Mathiowetz V, Volland G, Kashman N, Weber K. Adult norms for the Box and Block Test of manual dexterity. Am J Occup Ther. 1985 Jun;39(6):386-91. doi: 10.5014/ajot.39.6.386. PMID 3160243